CLINICAL TRIAL: NCT02139761
Title: L-tetrahydropalmatine (l-THP) Treatment for Cocaine Use Disorder
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study funding has not been established
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Deanna Kelly, Deanna L. Kelly Pharm.D., BCPP, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00059193
Record Dates: First submitted 2014-04-24; First posted 2014-05-15 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Cocaine Use
Keywords: Cocaine; Treatment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- l-tetrahydropalmatine (l-THP) (Active Comparator): Subjects will be dosed 30 mg BID (2 capsules total a day, total of 60mg/day), matching placebo or l-THP) (total 60 mg daily). The half-life of l-THP is about 10 hours, so subjects will reach steady state in about 2-3 days. The l-THP will be prepared at the University of Maryland School of Pharmacy to Chemistry under Good Manufacturing Practice (GMP) and standards. The identical placebo and active capsules will be manufactured and sent to the Maryland Psychiatric Research Center Pharmacy, where they will be stored, randomized and dispensed. Medication will be transported by the study staff to the participant once dispensing occurs.
  Interventions: Drug: l-tetrahydropalmatine (l-THP)
- Placebo (Placebo Comparator): Subjects will be dosed 30 mg BID (2 capsules total a day, total of 60mg/day), matching placebo or l-THP) (total 60 mg daily). The half-life of l-THP is about 10 hours, so subjects will reach steady state in about 2-3 days. The l-THP will be prepared at the University of Maryland School of Pharmacy to Chemistry under Good Manufacturing Practice (GMP) and standards. The identical placebo and active capsules will be manufactured and sent to the Maryland Psychiatric Research Center Pharmacy, where they will be stored, randomized and dispensed. Medication will be transported by the study staff to the participant once dispensing occurs.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: l-tetrahydropalmatine (l-THP) — Subjects will be dosed 30 mg BID (2 capsules total a day, total of 60mg/day), matching placebo or l-THP) (total 60 mg daily). The half-life of l-THP is about 10 hours, so subjects will reach steady state in about 2-3 days. The l-THP will be prepared at the University of Maryland School of Pharmacy to Chemistry under Good Manufacturing Practice (GMP) and standards. The identical placebo and active capsules will be manufactured and sent to the Maryland Psychiatric Research Center Pharmacy, where they will be stored, randomized and dispensed. Medication will be transported by the study staff to the participant once dispensing occurs.
  Arms: l-tetrahydropalmatine (l-THP)
Drug: Placebo — Subjects will be dosed 30 mg BID (2 capsules total a day, total of 60mg/day), matching placebo or l-THP) (total 60 mg daily). The half-life of l-THP is about 10 hours, so subjects will reach steady state in about 2-3 days. The l-THP will be prepared at the University of Maryland School of Pharmacy to Chemistry under Good Manufacturing Practice (GMP) and standards. The identical placebo and active capsules will be manufactured and sent to the Maryland Psychiatric Research Center Pharmacy, where they will be stored, randomized and dispensed. Medication will be transported by the study staff to the participant once dispensing occurs.
  Arms: Placebo

SUMMARY:
Cocaine continues to be one of the most widely used substances of abuse around the world. In the US, an estimated 1.4 million individuals (0.5%) > 12 years were current (past month) cocaine users in 2011. Currently, no FDA-approved pharmacologic treatments are available for cocaine addiction; thus, this remains a serious public health problem without an effective pharmacological treatment. A promising lead towards an effective treatment comes from a recent finding that pretreatment with oral l-tetrahydropalmitine (l-THP) in rats attenuated the cocaine seeking associated with a cocaine challenge, while having no motor effects. This finding stimulated our group to test the pharmacokinetics and safety of l-THP in a phase I study of people with cocaine use. Preliminary findings show l-THP is safe and well tolerated in cocaine users, with no adverse interactions with cocaine.

This study will test the efficacy and safety of l-THP for abstinence in those with cocaine addiction in a phase II pilot study (N=24). Secondarily, we will examine the effects of these medications on craving.

ELIGIBILITY:
Inclusion Criteria:

* men or non-pregnant/non-nursing women between the ages of 18 and 50 years
* meeting criteria for DSM-5 cocaine use disorder
* self-reported cocaine use (intranasal, IV or smoked) averaging at least weekly for the prior six months positive urine drug test for cocaine in the prior month
* HIV seronegative
* EKG without clinically significant abnormality
* normal blood pressure (systolic: 90-140 mmHg; diastolic: 50-90 mmHg) and resting heart rate (60-90 bpm)
* ability to adhere to the study restrictions and examination schedule
* women with reproductive potential must agree to the use of one of the following birth control methods (oral contraceptives, condom with spermicide, diaphragm, or intrauterine device) during the study and for 2 weeks after last medication dose.

Exclusion Criteria:

* participation in any investigational drug trial or clinical drug trial within 45 days before study entry
* history of clinically significant adverse reaction or hypersensitivity to cocaine or l-THP
* inability to communicate or co-operate with the investigators
* currently taking any prescribed psychoactive medication, e.g., anti- depressant, anti-psychotic, or mood stabilizer
* current clinically significant medical problem that might interfere with safe study participation. This includes pheochromocytoma, untreated hyperthyroidism, dehydration, fever, coronary artery disease, uncorrected congenital heart defect, seizures, electrolyte imbalance, uncontrolled diabetes mellitus, porphyria variegate, superventricular tachycardia, atrial fibrillation, cardiomyopathy, or uncontrolled hypertension.
* current Axis I Major Depression, Schizophrenia, or Bipolar Disorder.
* score below 10/12 on the Evaluation to Sign Consent (ESC)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
We will assess abstinence to cocaine as the outcome | 8 Weeks
  We will measure cocaine and its metabolite by urine drug test to assess for abstinence.

CONTACTS AND LOCATIONS:
Overall Officials: Deanna L Kelly, Pharm.D, BCPP, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Maryland Psychiatric Research Center, Catonsville, Maryland, United States